CLINICAL TRIAL: NCT07322549
Title: Amoxicillin/Clavulanic Acid Susceptibility in Acute Community-acquired Pneumonia Documented With Streptococcus Pneumoniae, Haemophilus Influenzae, or Staphylococcus Aureus Requiring Intensive Care Management: a Single-center Retrospective Study.
Brief Title: Amoxicillin/Clavulanic Acid Susceptibility in Acute Community-acquired Pneumonia Requiring Intensive Care Management
Acronym: CAP-ICU
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Other Study IDs: C-2025-006-MC
Record Dates: First submitted 2025-12-01; First posted 2026-01-07 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Severe Community-acquired Pneumonia
Keywords: Community-acquired pneumonia; Community-asquired aspiration pneumonia; Intensive care; Streptococcus pneumoniæ; Haemophilus influenzae; Staphylococcus aureus
MeSH Terms: conditions — Community-Acquired Pneumonia; Haemophilus Infections; Staphylococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with severe community-acquired pneumonia: Pneumonia documented with Streptococcus pneumoniae, and/or Haemophilus influenzae, and/or Staphylococcus aureus
  Interventions: Other: Susceptibility to AMC; Other: Susceptibilty to 3GC

INTERVENTIONS:
Other: Susceptibility to AMC — Susceptibility to AMC
Other: Susceptibilty to 3GC — Susceptibilty to 3GC

SUMMARY:
Severe community-acquired pneumonia (CAP) and community-acquired aspiration pneumonia (CAAP) are common reasons for adult emergency department visits and subsequent admission to the intensive care unit (ICU). Three bacteria are primarily implicated in this type of pneumonia: Streptococcus pneumoniae, Haemophilus influenzae, and Staphylococcus aureus.

Empirical antibiotic therapy for this condition is currently based on the use of beta-lactams. While third-generation cephalosporins (3GC) remain the beta-lactam of choice in French guidelines for CAP, the combination of Amoxicillin/Clavulanic Acid (AMC) at high-dose (>3g/day) could represent an alternative. AMC is already recommended for severe CAAP and for non-severe CAP in France, and for severe CAP in the UK and the United States. Furthermore, good practice guidelines encourage the use of empirical antibiotic therapies that are then subsequently tailored to the narrowest-spectrum agents based on antibiograms. This approach aims to limit the emergence of multidrug-resistant bacteria and reduce the risk of Clostridioides difficile colitis, which can increase patient morbidity and mortality.

This study aims to evaluate the susceptibility to AMC and 3GC, and to describe the empirical antibiotic therapies used and their subsequent adjustments, in adult patients admitted to the ICU for severe CAP and CAAP documented with Streptococcus pneumoniae, and/or Haemophilus influenzae, and/or Staphylococcus aureus.

DETAILED DESCRIPTION:
Observational retrospective monocentric cohort including all the consecutive adult ICU patients admitted from january 2018 to november 2022 with a CAP or a CAAP documented to Streptococcus pneumoniae, and/or Haemophilus influenzae, and/or Staphylococcus aureus.

ELIGIBILITY:
Inclusion Criteria:

1. Patient admitted to the ICU at Sainte-Musse Hospital between January 2018 and December 2022.
2. Diagnosis of severe CAP or CAAP within 48 hours of hospital admission, documented with Streptococcus pneumoniae, and/or Haemophilus influenzae, and/or Staphylococcus aureus (confirmed by blood culture and/or a respiratory sample), with an available antibiogram.

Exclusion Criteria:

1. Patient under 18 years old.
2. Patient hospitalized within 3 months prior to hospital admission.
3. Infectious documentation of another pathogen within 48 hours of hospital admission.
4. Nosocomial pneumonia.
5. Patient under legal guardianship (inmate, legal ward, curatorship).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU at Sainte-Musse Hospital between January 2018 and December 2022 with a diagnosis of severe CAP or CAAP
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Susceptibility rate to AMC and/or 3GC for identified bacteria at CAP or CAAP diagnosis | Up to 28 days
  The antibiotics of interest are:
  * The combination of Amoxicillin/Clavulanic Acid (AMC)
  * Third-generation cephalosporins (3GCs)

SECONDARY OUTCOMES:
Patient characteristics according to AMC sensitivity | Up to 28 days
  Comparison of patients' characteristics (chronic disease, ICU parameters) according to CAP with a documented bacteria susceptible to AMC or not.
Susceptibility rate to empirical recommended beta lactam (AMC, 3GC, and piperacillin/tazobactam) | Up to 28 days
  The rates of antibiotic use will be analyzed according to the following criteria:
  * Inappropriate: Inappropriate antibiotic spectrum.
  * Appropriate: Antibiotic spectrum appropriate for the identified pathogen.
  * Unjustified: Overly broad antibiotic spectrum.
Mortality rate | Up to 28 days
  Mortality at ICU discharge will be assessed overall and stratified by the appropriateness of antibiotic therapy (classified as inappropriate, appropriate, or unjustified).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Intercommunal Toulon La Seyne sur Mer, Toulon, Var, France